CLINICAL TRIAL: NCT00253474
Title: A Phase I Trial of Peginterferon Alfa-2b (PEG-Intron) for Plexiform Neurofibromas
Brief Title: PEG-Interferon Alfa-2b in Treating Young Patients With Plexiform Neurofibroma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 050232; 05-C-0232; NCI-P6670; CDR0000448811; NCT00156754 (obsolete NCT alias)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Neoplasm of Uncertain Malignant Potential; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: neoplasm of uncertain malignant potential; unspecified childhood solid tumor, protocol specific
MeSH Terms: interventions — peginterferon alfa-2a

INTERVENTIONS:
Biological: PEG-interferon alfa-2a

SUMMARY:
RATIONALE: PEG-interferon alfa-2b may interfere with the growth of tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of PEG-interferon alfa-2b in treating young patients with plexiform neurofibroma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of PEG-interferon alfa-2b in patients with unresectable plexiform neurofibroma. (Dose escalation portion of study closed to accrual as of 2/2005.)
* Determine the toxicity profile of this drug in these patients.

Secondary

* Obtain, preliminary, information about the efficacy of this drug in these patients.
* Evaluate the growth rate of plexiform neurofibroma using volumetric MRI analysis in patients treated with this drug.
* Evaluate the impact of this drug, in terms of "worst symptom" score, in these patients.

OUTLINE: This is a dose-escalation, multicenter study. (Dose-escalation portion of the study closed to accrual as of 2/2005.)

Patients receive PEG-interferon alfa-2b subcutaneously once weekly for 2 years in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of PEG-interferon alfa-2b until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 6 patients experience dose-limiting toxicity. A total of 12 patients receive treatment at the MTD.

After completion of study treatment, patients are followed every 6 months.

PROJECTED ACCRUAL: A total of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of plexiform neurofibroma which is progressive, symptomatic, or life threatening and for which there is no other standard medical management or surgical option
* Histologic confirmation of tumor is not required in the presence of consistent clinical and radiographic findings provided the following are true:

  * No clinical observation or scan suggestive of malignant transformation
  * Meets ≥ 1 of the following diagnostic criteria for neurofibroma type 1 (NF1):

    * Six or more cafe-au-lait spots (> 0.5 cm in prepubertal patients or > 1.5 cm in post pubertal patients)
    * Freckling in axilla or groin
    * Optic glioma
    * Two or more Lisch nodules
    * A distinctive bony lesion (e.g., dysplasia of the sphenoid bone, dysplasia, or thinning of long bone cortex)
    * A first degree relative with NF1
* No history of malignant peripheral nerve sheath tumor
* No active visual pathway glioma
* No active brain tumor or brain metastases

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* At least 12 months

Hematopoietic

* Absolute neutrophil count > 1,500/mm^3
* Hemoglobin > 10 g/dL
* Platelet count > 100,000/mm^3

Hepatic

* Bilirubin < 1.5 mg/dL
* SGPT ≤ 2 times upper limit of normal
* No significant hepatic dysfunction

Renal

* Creatinine based on age as follows:

  * ≤ 0.8 mg/dL (for patients age 5 years and under)
  * ≤ 1.0 mg/dL (for patients age 6 to 10 years)
  * ≤ 1.2 mg/dL (for patients age 11 to 15 years)
  * ≤ 1.5 mg/dL (for patients age 16 to 21 years) OR
* Creatinine clearance ≥ 70 mL/min

Cardiovascular

* No significant cardiac dysfunction
* No severe cardiovascular disease
* No cardiac arrhythmia requiring chronic treatment
* No congestive heart failure
* No symptomatic ischemic heart disease

Pulmonary

* No significant pulmonary dysfunction

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No serious infection
* No other significant unrelated systemic illness
* No significant organ dysfunction
* No other malignancy except surgically cured nonmelanoma skin cancer or carcinoma in situ of the cervix
* No history of severe psychiatric condition or psychiatric disorder requiring hospitalization
* No history of suicidal ideation or attempt
* No thyroid dysfunction unresponsive to therapy
* No uncontrolled diabetes mellitus
* No history of HIV positivity
* No alcohol or drug abuse

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy
* No concurrent colony-stimulating factors (e.g., erythropoietin or filgrastim [G-CSF])

Chemotherapy

* No concurrent chemotherapy for this disease

Endocrine therapy

* No concurrent chronic systemic corticosteroids
* No concurrent hormonal therapy for this disease

Radiotherapy

* No concurrent radiotherapy for this disease

Surgery

* Prior surgery allowed provided it has been at least 21 days since surgery and there is presence of residual tumor

Other

* Recovered from prior therapy
* More than 30 days since prior investigational agents

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2005-09; Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C. Widemann, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- United States (4):
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Result] Jakacki RI, Dombi E, Potter DM, Goldman S, Allen JC, Pollack IF, Widemann BC. Phase I trial of pegylated interferon-alpha-2b in young patients with plexiform neurofibromas. Neurology. 2011 Jan 18;76(3):265-72. doi: 10.1212/WNL.0b013e318207b031. PMID 21242495